CLINICAL TRIAL: NCT02722512
Title: A Phase I and Feasibility Trial of Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine for Pediatric Patients With Newly Diagnosed Intracranial High Grade Glioma and Recurrent Resectable Intracranial High Grade Glioma and Ependymoma
Brief Title: Trial of Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of substantial evidence for immune responses in response to vaccination.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Angela Waanders, Section Head, Pediatric NeuroOncology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-362
Record Dates: First submitted 2016-03-17; First posted 2016-03-30 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma Multiforme; Astrocytoma, Grade III; Anaplastic Ependymoma; Clear Cell Ependymoma; Ependymoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Ependymoma | interventions — vitespin; Transurethral Resection of Bladder; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Newly Diagnosed High Grade Glioma (HGG) (Experimental): Heat Shock Protein Peptide Complex-96 (HSPPC-96) therapy will be given between 0-28 days after the completion of radiation therapy (XRT) AND no more than 60 days from completion of XRT. Vaccine will be given once weekly for 4 weeks. The 4 weeks (28 days) of vaccine administration will be followed by an observation visit. In patients with sufficient vaccine (on both Arms A and B), a maintenance therapy will be instituted. It will be administered at the same dose the patient was enrolled at and given every 2 weeks until vaccine is exhausted or there is evidence of tumor progression. The first dose of maintenance vaccine should be administered 7 days after completion of the observation visit.
  Interventions: Biological: Heat Shock Protein Peptide Complex-96 (HSPPC-96); Procedure: Tumor Resection; Radiation: Radiation
- Recurrent HGG and Ependymoma (Experimental): On Arm B, Heat Shock Protein Peptide Complex-96 (HSPPC-96) will be given as soon as possible after tumor resection post-operative recovery and sufficient time for vaccine preparation (typically 0-28 days post-operatively) AND no more than 60 days post-operatively. Vaccine will be given once weekly for 4 weeks. These 4 weeks (28 days) of vaccines will be followed by an observation visit. In patients with sufficient vaccine, a maintenance therapy will be given. It will be given at the same dose the patient was enrolled at and given every 2 weeks until vaccine is exhausted or there is evidence of tumor progression. The first dose of maintenance vaccine should be given 7 days after completion of the observation visit.
  Interventions: Biological: Heat Shock Protein Peptide Complex-96 (HSPPC-96); Procedure: Tumor Resection

INTERVENTIONS:
Biological: Heat Shock Protein Peptide Complex-96 (HSPPC-96) — The vaccine is patient specific, created from the patient's own brain tumor resected at a clinically necessary surgery. The vaccine is administered intradermally on a weekly basis.
Procedure: Tumor Resection — Clinically-indicated removal of the tumor
Radiation: Radiation — Focal Radiation Therapy
  Arms: Newly Diagnosed High Grade Glioma (HGG)

SUMMARY:
The purpose of this study is to determine whether Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine is an feasible and safe treatment for pediatric patients with newly-diagnosed High-Grade Gliomas or recurrent, resectable High-Grade Gliomas and Ependymomas.

DETAILED DESCRIPTION:
Immunotherapy for Brain Tumors:

Although it is usually ineffective alone, it has long been recognized that the immune system of tumor bearing hosts (human and animal models) does, indeed, mount an endogenous immune-mediated response to tumor. Unfortunately, this immune response alone is not sufficient in combating tumor. The balance of immune response and immune regulation often mitigates this anti-tumor response. Several mechanisms within tumor-bearing hosts compromise the efficacy of this anti-tumor immune response, including low levels of expression of co-stimulatory molecules such as the B7 family of immune-regulatory ligands, the tumor's local production of immunosuppressive factors and the tumor's ability to over-express pro-survival factors thus escaping destruction by the host immune system. However, many have hypothesized that if this immune response can be better harnessed and/or magnified, there is potential for heightened tumor responses.

A number of specific observations support the use of immunotherapy to treat brain tumors. Data published supports a possible correlation between HIV mediated immunosuppression and the development of intracranial glial tumors. Immunosuppression in transplant recipients has also been implicated in the development of intracranial glioma. Further supporting this hypothesis are documented rare cases of long-term remission of malignant brain tumors following significant post-operative infection. These observations have fueled the idea that a heightened immune system may confer some protection against intracranial tumors. With this in mind, one hypothesis is that successful active immunotherapy for patients with brain tumors will require development of a specific peptide or polyvalent vaccines in an effort to further stimulate the host's immune system against specific tumor-associated antigens.

It has been well established that mice can be immunized against syngeneic tumors. Heat shock protein-peptide complexes isolated from a specific tumor can been utilized to elicit both prophylactic and therapeutic immunity against the specific cancer from which the preparations have been isolated. Overexpression of heat shock protein-chaperone complexes (HSPPC) in brain tumor cells suggests that HSPPC are a meaningful target antigen for a brain tumor vaccine. Moreover, in addition to generating tumor-specific immunity, vaccination with heat shock protein peptide complexes in animal models generates therapeutic responses. Since an immune response has not been widely evaluated for pediatric brain tumors, this study will test the safety and feasibility of producing and administering a vaccine capable of generating an autologous, anti-tumor immune response.

HSPPC-96:

Heat shock proteins are up-regulated along with tissue-specific chaperone peptides in the setting of cellular stress to prevent damage and aggregation of the proteome. Therefore, heat shock protein peptide complexes (HSPPC) provide a cytoprotective effect. Overexpression of heat shock proteins has been described in malignant glioma and medulloblastoma cells. HSPPC-96 is an autologous tumor-derived vaccine that has been under clinical investigation for the treatment of a variety of cancer types, including adult high-grade glioma (HGG). It is composed of the 96-kilodalton (KDa) heat shock protein, glycoprotein 96 (gp96), attached to autologous tumor-derived peptides. The gp96 glycoprotein in HSPPC-96 is a highly conserved, abundant, non-polymorphic stress protein found in every cell type of the body. Gp96 isolated from normal or tumor tissues is found in complex with peptides that are specific to the original tissue. Mouse models have shown that HSPPC-96 confers protective immunity only to the tumor from which it is derived and not to genetically distinct tumors or normal tissue.

When injected into the host, HSPPC-96 interacts with antigen presenting cells (APCs) via specific receptors. Once internalized by the APCs, the peptides chaperoned by the HSP are transferred to major histocompatibility complex (MHC) class I and class II molecules in intracellular compartments and eventually expressed at the cell surface. T-cells then recognize the MHC-peptide complexes and are stimulated. HSP-peptide complexes are unique in their ability to elicit an antigen-specific cytotoxic T-cell response. Additionally, cluster of differentiation 4 (CD4+) T cells and natural killer (NK) cells are also recruited adding to the tumor-associated immunity.

Some advantages of heat shock protein-peptide vaccines for immunotherapy are that it elicits a cluster of differentiation (CD8+) T cell response in spite of exogenous administration, it circumvents the need for identification of T-cell epitopes of individual cancers, and it minimizes the possibility of generating epitope variants. Furthermore, heat shock protein-peptide complexes have elicited tumor rejection and CD8+ T cell response without adjuvant therapies. Heat shock protein-peptide complexes, such as HSPPC-96, can be isolated from human tumors, and when injected back into the patient from whom they were isolated, may present a unique opportunity to deliver a vaccine specific to that patient.

ELIGIBILITY:
Inclusion Criteria:

* Arm A: Newly Diagnosed High Grade Glioma Tumor
* Arm B: Recurrent, resectable High Grade Glioma or Ependymoma
* Stable Neurologic Status
* Lanksy/Karnofsky score greater than or equal to 50.
* Adequate Bone Marrow Function (ANC≥ 1000/μL, platelets≥ 100,000/μL transfusion independent, Hemoglobin ≥ 8.0 gm/dL with or without transfusion support)
* Adequate Liver Function (Bilirubin ≤ 2x institutional normal for age, Alanine transaminase (ALT) ≤ 5x institutional normal for age, Aspartate Aminotransferase (AST) ≤ 5x institutional normal for age)
* Adequate Renal Function (Normal creatinine for age and/or glomerular filtration rate ≥ 70 mls/min/1.73 m2)
* Female patients of childbearing potential must have a negative serum or urine pregnancy test

Exclusion Criteria:

* Patients with unresectable disease are not eligible.
* Patients with primary spinal cord tumors are not eligible.
* Patients with metastatic disease are not eligible for Arm A (this does NOT apply to Arm B).
* Patients with a known allergy to any component of the vaccine or any compounds of similar chemical or biologic composition of the vaccine are not eligible.
* Patients with known auto-immune disease are excluded.
* Patients with known immunodeficiency are excluded.
* Patients with a concurrent malignancy are excluded.
* Clinically Significant Concurrent Illness
* Patients receiving any other anticancer or investigational drug
* Patients with uncontrolled seizure disorders
* Patients whose central nervous system (CNS) tumor is considered a secondary malignancy from prior therapies

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
The rolling 6 statistical design will be utilized to establish the MTD and RP2D of HSPCC autologous vaccine in children with newly diagnosed high grade glioma (HGG) following focal radiation therapy and in recurrent HGG and ependymoma given alone. | 36 months

SECONDARY OUTCOMES:
To estimate the progression-free survival distribution in children with recurrent and resectable HGG treated with HSPPC-96 vaccine therapy alone (Arm B). | 60 months
To estimate the progression-free survival distribution in children with recurrent and resectable ependymoma treated with HSPPC-96 vaccine therapy alone (Arm B). | 60 months
To evaluate patient immune responses as measured by immune correlates in the above patient groups. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided